CLINICAL TRIAL: NCT03513601
Title: Treatment of Elderly Patients With Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2017-10
Record Dates: First submitted 2017-10-31; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Curative effect evaluation; Adverse reactions; Clinical characteristics; PR; PFS; OS
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- (R)-CHOP regimen (Experimental): (R)-CHOP regimen((rituximab)，cyclophosphamide，epirubicin，vincristine and prednisone)，(rituximab 375mg/m2 d0 ivgtt),cyclophosphamide 750mg/m2 d1、8 ivgtt,epirubicin 50mg/m2 d1、8 ivgtt,vincristine 2mg d1、8 ivgtt,prednisone 60mg d1-5 po.Every 21 days for one cycle and six cycles are required. Efficacy was evaluated every two cycles.
  Interventions: Drug: (R)-CHOP regimen
- (R)-CVP regimen (Experimental): (R)-CVP regimen((rituximab)，cyclophosphamide，vincristine and prednisone) The dose of the chemical was reduced by 20%，(rituximab 375mg/m2 d0 ivgtt),cyclophosphamide 750mg/m2 d1、8 ivgtt,vincristine 2mg d1、8 ivgtt,prednisone 60mg d1-5 po.Every 21 days for one cycle and one or two cycles are required. Efficacy was evaluated every two cycles. Subsequent (rituximab 375mg/m2 d0 ivgtt)， oral cyclophosphamide .
  Interventions: Drug: (R)-CVP regimen

INTERVENTIONS:
Drug: (R)-CHOP regimen — (rituximab 375mg/m2 d0 ivgtt),cyclophosphamide 750mg/m2 d1、8 ivgtt,epirubicin 50mg/m2 d1、8 ivgtt,vincristine 2mg d1、8 ivgtt,prednisone 60mg d1-5 po.Every 21 days for one cycle and six cycles are required. Efficacy was evaluated every two cycles.
  Other Names: (rituximab)，CTX，VCR，EPI，PDN
  Arms: (R)-CHOP regimen
Drug: (R)-CVP regimen — The dose of the chemical was reduced by 20%，(rituximab 375mg/m2 d0 ivgtt),cyclophosphamide 750mg/m2 d1、8 ivgtt,vincristine 2mg d1、8 ivgtt,prednisone 60mg d1-5 po.Every 21 days for one cycle and one or two cycles are required. Efficacy was evaluated every two cycles. Subsequent (rituximab 375mg/m2 d0 ivgtt)， oral cyclophosphamide .
  Other Names: (rituximab)，CTX，VCR，PDN,20 percent reduction in chemical therapy
  Arms: (R)-CVP regimen

SUMMARY:
To explore the clinical features and efficacy evaluation of large b-cell lymphoma in old age.

DETAILED DESCRIPTION:
The results of the analysis of the treatment of large b-cell lymphoma in old age were analyzed, and the treatment of large B cell lymphoma was provided.

ELIGIBILITY:
Inclusion Criteria:

* Above 70 years old，Pathology proved to be diffuse large B cell lymphoma，Estimated survival time > 3 months，None of chemotherapy contraindication;At least one measurable lesion according to RECIST;None of other serious diseases;Patients could be followed up;None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.

volunteers who signed informed consent.

Exclusion Criteria:

* Currently undergoing chemotherapy, radiotherapy and targeted therapy (received chemotherapy within 3 weeks, received radiotherapy within 2 weeks, or has not recovered from any previous treatment of acute toxicity);Patients with uncontrolled medical problems (including active infection, uncontrolled diabetes, severe heart, liver, kidney dysfunction and interstitial pneumonia, etc.); Pregnant or lactating women;Serious medical illness likely to interfere with participation;Chemotherapy contraindication such as cachexia; patients with other malignancies previously;Serious infection;The evidence of peripheral nervous disorder or dysphrenia; patients estimated to be unsuitable by investigator.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase(approximately 24 months)
  Progression-free survival

SECONDARY OUTCOMES:
overall survival | up to the date of death (approximately 5 years)
  overall survival
disease control rate | every 6 weeks,up to completion of treatment(approximately 18 weeks )]
  disease control rate
objective remission rate | every 6 weeks,up to completion of treatment(approximately 18 weeks )]
  objective remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China